CLINICAL TRIAL: NCT01936974
Title: Platinum-Gemcitabine-Avastin (PGA) for Platinum-resistant/Refractory, Paclitaxel-Pretreated Recurrent Ovarian and Peritoneal Carcinoma
Brief Title: (PGA) for Platinum-resistant/Refractory, Paclitaxel-Pretreated Recurrent Ovarian and Peritoneal Carcinoma
Acronym: PGA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-27
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Carcinoma; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Gemcitabine; Bevacizumab; Carboplatin; Cisplatin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platinum, Gemcitabine and Bevacizumab (Experimental): Platinum:
  1. Carboplatin* on day 1
     *If a patient is allergic to carboplatin, then give
  2. Cisplatin** on day 1
     **If a patient is allergic to cisplatin and carboplatin, then give
  3. Oxaliplatin on day 1
  Gemcitabine on day 1 only
  Bevacizumab on day 1
  Interventions: Drug: Gemcitabine; Drug: Bevacizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Oxaliplatin
- Gemcitabine and Bevacizumab (Active Comparator): Gemcitabine on days 1 and 8
  Bevacizumab on day 1
  Interventions: Drug: Gemcitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine — Patient to receive gemzar
  Other Names: Gemzar
Drug: Bevacizumab — Patient to receive avastin
  Other Names: Avastin
Drug: Carboplatin — Patient to receive carboplatin
  Other Names: Paraplatin
  Arms: Platinum, Gemcitabine and Bevacizumab
Drug: Cisplatin — Patient to receive cisplatin
  Other Names: Platinol
  Arms: Platinum, Gemcitabine and Bevacizumab
Drug: Oxaliplatin — Patient to receive Oxaliplatin
  Other Names: Eloxatin
  Arms: Platinum, Gemcitabine and Bevacizumab

SUMMARY:
To evaluate progression-free survival with two chemotherapy regimens on platinum-resistant/refractory ovarian and peritoneal carcinoma

DETAILED DESCRIPTION:
This study will evaluate progression-free survival (PFS)for the regimen of gemcitabine and bevacizumab with or without a platinum agent on platinum-resistant/refractory ovarian and peritoneal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with histologically confirmed, recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer
2. Disease progression during or within 6 months of previous platinum-based chemotherapy including the following 4 categories:

   1. Primary platinum-refractory: Previously untreated patients who do not achieve at least a partial response to platinum-based chemotherapy
   2. Primary platinum-resistant: Previously untreated patients who have achieved at least a partial response to platinum-based chemotherapy but experience a relapse within a period of 6 months of its conclusion
   3. Secondary platinum-refractory: Previously treated patients have a relapse 6 months after the conclusion of chemotherapy, but fail to achieve at least a partial response
   4. Secondary platinum-resistant: Previously treated patients have a relapse 6 months after the conclusion of chemotherapy, achieve at least a partial response with platinum-based therapy as 2nd-line therapy, but experience relapse within 6 months
3. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2 and a life expectancy >3 months.
4. Absolute neutrophil count > 1500 mm^3, platelet count ≥ 100×10^9 L, hemoglobin ≥ 8.5 g/dL
5. Serum creatinine ≤1.5 times the upper limit of the normal range, total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 5 times the upper limit of normal range
6. No remaining grade 2 or higher toxicity from prior cancer therapies unless judged to be clinically insignificant by the Principal Investigator
7. At least three (3) weeks from prior chemotherapy

Exclusion Criteria:

1. Inadequate renal function with a calculated creatinine clearance less than 51 mL/min
2. Uncontrolled cardiac disease, congestive heart failure, angina, or hypertension
3. Myocardial infarction or unstable angina within 2 months of treatment
4. Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B or C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol)
5. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks, pulmonary embolism within the past 6 months
6. Bleeding diathesis or significant coagulopathy
7. Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug
8. Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug
9. History of fistula, GI perforation, or intrabdominal abscess
10. Serious non-healing wound, ulcer, or bone fracture
11. clinical signs or symptoms of GI obstruction and/or requirement for parenteral hydration or nutrition
12. Known CNS disease except for treated brain metastasis
13. Known platinum drug allergy
14. Prior treatment with Platinum + Gemcitabine + Avastin, Gemcitabine + Avastin or Gemcitabine alone
15. Prior treatment with more than three (3) lines of chemotherapy including adjuvant chemotherapy
16. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
17. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
18. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Platinum, Gemcitabine and Bevacizumab: Platinum:
  1. Carboplatin* on day 1
     *If a patient is allergic to carboplatin, then give
  2. Cisplatin** on day 1
     **If a patient is allergic to cisplatin and carboplatin, then give
  3. Oxaliplatin on day 1
  Gemcitabine on day 1 only
  Bevacizumab on day 1
  Gemcitabine
  Bevacizumab
  Carboplatin
  Cisplatin
  Oxaliplatin
- Gemcitabine and Bevacizumab: Gemcitabine on days 1 and 8
  Bevacizumab on day 1
  Gemcitabine
  Bevacizumab
Period: Overall Study
Arm/Group | Platinum, Gemcitabine and Bevacizumab | Gemcitabine and Bevacizumab
Started | 2 | 5
Completed | 0 | 0
Not Completed | 2 | 5
Not completed — Physician Decision | 2 | 5

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected. No data was collected for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum, Gemcitabine and Bevacizumab | Gemcitabine and Bevacizumab | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Evaluate progression-free survival between the two regimens.
Time Frame: One Year
Population: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information.After much effort, results were not able to be retained.
Arm/Group | Platinum, Gemcitabine and Bevacizumab | Gemcitabine and Bevacizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Description: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Arm/Group | Platinum, Gemcitabine and Bevacizumab | Gemcitabine and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes